CLINICAL TRIAL: NCT00473707
Title: A Randomized Trial of Active Versus Expectant Management of the Third Stage of Labor
Brief Title: Active Versus Expectant Management of the Third Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Danielle Castagnola, Christiana Care Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26008
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Postpartum Hemorrhage
Keywords: Third stage of labor
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Active management of the third stage of labor- oxytocin infusion after delivery of fetus, gentle cord traction, and fundal massage
  Interventions: Procedure: Active management of the third stage of labor; Drug: Oxytocin and gentle cord traction with fundal massage
- 2 (Other): Expectant management of the third stage of labor
  Interventions: Procedure: Expectant management of the third stage of labor; Drug: Oxytocin

INTERVENTIONS:
Procedure: Active management of the third stage of labor — standardized oxytocin infusion (10 units of oxytocin in 500 mL of Ringers lactate over 20 minutes) immediately following delivery of the fetus with gentle cord traction and fundal massage
  Arms: 1
Procedure: Expectant management of the third stage of labor — standardized oxytocin infusion (10 units of oxytocin in 500 mL of Ringers lactate over 20 minutes) in combination with maternal expulsion efforts once spontaneous separation of the placenta had begun
  Arms: 2
Drug: Oxytocin and gentle cord traction with fundal massage — standardized oxytocin infusion (10 units of oxytocin in 500 mL of Ringers lactate over 20 minutes) immediately following delivery of the fetus with gentle cord traction and fundal massage
  Arms: 1
Drug: Oxytocin — standardized oxytocin infusion (10 units of oxytocin in 500 mL of Ringers lactate over 20 minutes) in combination with maternal expulsion efforts once spontaneous separation of the placenta had begun
  Arms: 2

SUMMARY:
The purpose of this study is to determine if giving oxytocin immediately after delivery causes less bleeding, transfusion needs and hastens delivery of placenta.

DETAILED DESCRIPTION:
Postpartum hemorrhage is the leading cause of maternal mortality worldwide. During the third stage of labor, the period following the delivery of the baby until the delivery of the placenta, the patient is at increased risk for blood loss. Controversy remains as to the optimal method of delivering the placenta. Two predominant, yet very different, strategies have emerged. Expectant management is most commonly used in the United States. This includes waiting for signs of placental separation, followed by maternal pushing to expel the placenta. Then uterotonic agents are administered,usually oxytocin. This is in contrast to active management, which consists of uterotonic administration immediately following delivery of the fetus, in association with gentle umbilical cord traction and fundal massage. This is the predominant practice in the United Kingdom, where the uterotonic agents of choice are either oxytocin alone, or a combination of oxytocin and ergometrine.

Comparison: Active management with oxytocin to expectant management of the third stage of labor on the effect of postpartum hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Cephalic presentation
* >37 weeks gestation
* >16 years of age

Exclusion Criteria:

* Multiple gestation
* Breech presentation
* Blood dyscrasias
* Multiparous females Para >5
* Placenta previa
* Patients on anticoagulants
* Previous history of postpartum hemorrhage
* IUFD
* Non-reassuring fetal heart rate pattern

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2002-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Incidence of postpartum hemorrhage, defined as estimated blood loss (EBL) 500mL or greater | reported immediately after delivery

SECONDARY OUTCOMES:
Mean change in hematocrit from before delivery to the first postpartum day | 24 hours
Rate of maternal blood transfusion | 48 hours
Duration of the third stage of labor | 60 minutes
Incidence of retained placenta | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Castagnola, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States